CLINICAL TRIAL: NCT04283773
Title: Immunohistochemical Evaluation of Protein P16 Expression in Ovarian Germ Cell Tumors.
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar A Ahmed, Demonstrator at Pathology department - faculty of medicine - Assiut university., Assiut University
Other Study IDs: 17100871; 2019-09-05-001-R1 (Other Grant/Funding Number: Grant office - faculty of medicine - Assiut university)
Record Dates: First submitted 2020-02-23; First posted 2020-02-25 (Actual); Results first posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Ovarian Neoplasms; Germ Cell Tumors; Immunohistochemistry
Keywords: OGCTs, P16 , Ki67 , IHC
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms, Germ Cell and Embryonal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Formalin fixed paraffin embedded blocks of 62 ovarian specimens will be included in this study. These specimens will be divided into 2 groups:
  1-42 surgically resected ovarian germ cell tumors specimens: 22 malignant ones( dysgerminoma , immature teratoma and yolk sac tumor) as a case group and equal 20 benign ones (mature cystic teratoma ) as comparison group .
  2- 20 normally apparent ovaries that surgically resected with specimens of total abdominal hysterectomy and salpingo-Oopherctomy for non-ovarian causes in perimenopausal women as a control group .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Malignant ovarian germ cell tumors ( MOGCTs).: 22 cases of malignant ovarian germ cell tumors ; include Dysgerminoma , yolk sac tumor and immature teratomas will be treated by anti P16 antibody and Ki67 antibody.
  Interventions: Combination Product: p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267); Combination Product: Ki67 antibody (DAKO) for malignant cases only
- Mature cystic teratomas.: 20 cases of mature teratomas will be treated by anti P16 antibody .
  Interventions: Combination Product: p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267)
- Normally apparent ovaries.: 20 cases of normally apparent ovaries will be treated by anti P16 antibody .
  Interventions: Combination Product: p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267)

INTERVENTIONS:
Combination Product: p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267) — Treatment of slides that cut from paraffin embedded blocks related to groups by immunohistochemical method by p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267).
Combination Product: Ki67 antibody (DAKO) for malignant cases only — Treatment of slides that cut from paraffin embedded blocks related to malignant case group by immunohistochemical method by Ki67 antibody.
  Groups: Malignant ovarian germ cell tumors ( MOGCTs).

SUMMARY:
Ovarian germ cell tumors (OGCTs) constitute 10% of ovarian tumors in Egypt and mainly affect young females. Teratomas are the most common type.Most of teratomas is benign. However, it is liable for malignant transformation. Others are malignant including dysgerminoma, immature teratoma, yolk sac tumor,.etc and accounts 1-1.5% of cancers in young females. The pathogenesis of OGCTs is not clearly understood.

P16 is a member of cyclin-dependent kinase (CDK) inhibitors. It arrests the cell cycle in G1 phase, so it is known as a tumor suppressor protein.P16 immunohistochemical(IHC) expression has been widely investigated in different cancers. Its IHC expression is either absent or overexpressed. Overexpression of p16 is documented in Human Papilloma Virus related endocervical neoplasms and High grade squamous intraepithelial lesions of the vulvovaginal region.Absence of p16 expression is detected in multiple cancers such as Lung cancer, colorectal cancer and lymphoma.

P16 IHC expression in OGCTs is poorly investigated. One study suggests that absent p16 is involved in proliferation of malignant OGCTs via molecular assessment.Another study suggested that decrease P16 is involved in malignant transformation of Mature cystic teratoma to squamous cell carcinoma.However, Previous studies are still limited and recommended further studies to confirm its results.

As the role of altered P16 protein in OGCTs is not widely investigated, we hypothesized that abnormal P16 expression may be involved in its pathogenesis and germ stem cell proliferation.This will give more information about molecular pathways of germ stem cell proliferation to give a hope for CDK inhibitors as novel target therapies in the management of OGCTs.

DETAILED DESCRIPTION:
In this study , we aim to :

1-Evaluate the immunohistochemical expression of p16 in neoplastic component of benign and malignant OGCTs and scoring its immunoreactivity.

2-Correlate between P16 immunohistochemical expression in MOGCTs with Ki 67 proliferating index and FIGO staging.

1. Type of the study: Matched case-control study.
2. Study subjects:

   1. Inclusion criteria: Different types of Ovarian germ cell tumors including : benign ( mature cystic teratoma ) and malignant ones ( dysgerminoma , immature teratoma and yolk sac tumor ) .
   2. Exclusion criteria:

      Any criteria that not fulfill the inclusion criteria such as resected ovarian tumors other than ovarian germ cell tumors e.g epithelial ovarian tumors, sex cord -stromal tumors or metastatic ovarian lesions.
      * The study protocol was approved by the Institutional Review Board at Faculty of medicine, Assiut University in December, 2019 (IRB No.17100871) and Ethical approval for this study was obtained from the committee of medical ethics, Faculty of medicine, Assiut University.
      * Study Setting: IHC lab of Pathology department, Faculty of medicine, Assiut University.
      * Tissue sampling: Sixty-two formalin fixed ,paraffin wax-embedded ovarian specimens were obtained from departments of surgical pathology in Assiut University Hospital (AUH) and South Egypt cancer institute (SECI) from January 2010 to January 2021. These specimens includes:

      (Group A) 22 malignant ovarian germ cell tumors (MOGCTs), (Group B) 20 apparent normal ovarian tissue as a control group and (Group C) 20 mature cystic teratomas as equal benign comparison group.

      Group A constitutes 5 dysgerminomas, 8 immature teratomas (four of them Grade II and the other four are Grade III, FIGO grading system) and 9 yolk sac tumors. The patients ranged in age from 12 to 23 years (median age 16.5 years). The initial diagnosis of each MOGCTs was re-evaluated according to the WHO Classification of Ovarian Tumors.

      Group B includes normally apparent ovaries that surgically resected with specimens of total abdominal hysterectomy and salpingo-opherctomy for non-ovarian, non-malignant causes as multiple fibroid uterus and adenomyosis as a control group. The patients ranged in age from 42 to 64 years (median 50 years old).

      All available Hematoxylin and eosin stained slides were examined by two independent pathologists by routine light microscopy and the most representative one or two tissue blocks were used for immunohistochemical staining. The clinical and pathological data includes age, grade, stage, recurrence of lesions were evaluated according to pathological reports.
      * Immunohistochemistry: The tissue samples were formalin-fixed, paraffin embedded tissue blocks, and were stored at room temperature. Thin sections of 4 um thickness were cut from selected representative tissue blocks, and were taken on to coated slides, kept in an oven at 70-C for 25 minutes, deparaffinized by washing in two containers of xylene for 15 minutes for each and rehydrated through serial dilutions (100% , 90% , 80% , 70 %) of alcohol for 5 minutes in each dilution. Then, sections were treated by 3% Hydrogen peroxide for 10 minutes to prevent nonspecific background followed by PBS buffer wash 4 times adequately. For antigen retrieval, the slides were kept in citrate buffer (PH = 6) and autoclaved at 90-C for 15 minutes and left to cool to room temperature. The slides were washed with PBS buffer 4 times adequately and the tissue sections were incubated with primary antibody; p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267) (MA5-27905) at a dilution of 1:500 overnight, followed by incubation with secondary antibody; Polyvalent polymer-HRP for 10 minutes for each step followed by adequate 4 times of PBS buffer wash. The tissues were then treated with Diaminobenzidine chromogen (DAP-chromogen) for brown color development for 10 minutes. Then, sections were treated by Mayer hematoxylin as the counter stain for 2 minutes.

      For sections received from malignant cases only , we add additional Ki67 IHC staining as tissue sections after deparffinization and blocking by 3% hydrogen peroxidase were incubated with primary antibody; Ki67 antibody (DAKO), ready to use for 20 minutes, followed by incubation with secondary antibody; Polyvalent polymer-HRP for 20 minutes, followed treatment with Diaminobenzidine chromogen (DAP-chromogen) for brown color development for 5 minutes. Then, sections were treated by Mayer hematoxylin as the counter stain for 2 minutes.

      The slides were washed by tap water, dehydrated through serial dilutions of alcohol, washed by xylene for a short period, and mounted with DPX.

      The normal apparent ovarian tissues were used as controls. Sections from cervical non keratinized Squamous cell carcinoma with block p16 expression, were used as positive controls; and the tissue slides without the primary antibody treatment served as the negative controls.

      -Immunohistochemical evaluation: For P16 IHC staining, the percentage of P16 positive cells and the location of positive signals (nuclear or cytoplasmic) were visually estimated for neoplastic components of all lesions. German Semi-quantitative scoring system were used to evaluate P16 expression as every tumor will be given a score according to the intensity of the cytoplasmic and nucleic staining (no staining = 0, weak staining = 1, moderate staining = 2, strong staining = 3) And the extent of stained cells (0% = 0, 1-10% = 1, 11-50% =2, 51-80% = 3, 81-100% = 4). The final immunoreactive score will be determined by multiplying the intensity scores with the extent of positivity scores of stained cells, with the minimum score of 0 and a maximum score of 12 ( score 0, 1,2,3,4,6,8,9 and 12).

      For KI67 IHC staining for malignant cases only, percentage of nuclear positivity stained cells were assessed, regardless intensity of staining in all sections examined (at least 1000 tumor cells were counted per section for estimation of KI index).

      -Statistical analysis: Data were analysed using IBM-SPSS version 24. Numerical data were presented as mean and standard deviation, while categorical data were presented as number and percentage. Descriptive statistics: Means, standard deviations, medians, ranges, and percentages were calculated. Test of significances: for continuous variables with more than two categories; ANOVA test was calculated to test the mean differences of the data that follow normal distribution and independent sample Kruskal-Wallis was used to compare the median difference between groups that do not follow normal distribution, post-hoc test was calculated using Bonferroni corrections. Correlation analysis was used (Spearman' Ranked correlation, 2-tailed).

      A p-value < 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Ovarian germ cell tumors :

  1. 20 benign ( mature cystic teratoma ).
  2. 22 malignant ones ( 5 dysgerminoma , 8 immature teratoma and 9 yolk sac tumor).
  3. 20 Normal ovaries .

Exclusion Criteria:

1. Epithelial ovarian tumors
2. sex cord -stromal ovarian tumors.
3. metastatic ovarian lesions.

Ages: 6 Months to 1 Year | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: Sixty-two formalin-fixed, paraffin wax-embedded ovarian specimens .These specimens includes:
  (Group A) 22 malignant ovarian germ cell tumors (MOGCTs): 5 dysgerminomas, 8 immature teratomas (four of them Grade II and the other four are Grade III, FIGO grading system) and 9 yolk sac tumors. The patients ranged in age from 12 to 23 years (median age 16.5 years). The initial diagnosis was re-evaluated according to the WHO Classification of Ovarian Tumors.
  , (Group B) 20 apparent normal ovarian tissue as a control group that are surgically resected with TAH and salpingo-opherctomy for non-ovarian, non-malignant causes. The patients ranged in age from 42 to 64 years (median 50 years old).
  and(Group C) 20 mature cystic teratomas as equal benign comparison group.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-12-24 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Ahmed, Master, Principal Investigator — Pathology department- Faculty of medicine - Assiut university
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Clinical Study Report — https://journals.lww.com/greenjournal/Fulltext/2006/05000/Malignant_Germ_Cell_Tumors_of_the_Ovary.19.aspx — Incidence and Survival Rates for Female Malignant Germ Cell Tumors
- Available data/document: Clinical Study Report — https://synapse.koreamed.org/DOIx.php?id=10.3802/jgo.2012.23.2.125 — Early diagnosis of malignant-transformed ovarian mature cystic teratoma: fat-suppressed MRI findings

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 year .
Groups:
- IHC of P16 Expression in Malignant Ovarian Germ Cell Tumors.: 22 cases of malignant ovarian germ cell tumors ; 5cases of dysgerminoma ( one of them is bilateral) , 9 cases of yolk sac tumor and 8 cases of immature teratoma. These cases are treated by anti P16 antibody( p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267) , 1:500 concentration, over night duration and then treated by DAP secondary antibody . Finally assessed by visualized peroxidase method. and also treated by Ki67 antibody.
- IHC of P16 Expression in Benign Ovarian Germ Cell Tumors ( Mature Cystic Teratomas).: 20 cases of benign ovarian germ cell tumors ( Mature cystic teratomas). These cases are treated by anti P16 antibody( p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267) , 1:500 concentration, over night duration and then treated by DAP secondary antibody.
- IHC of P16 Expression in Normal Ovarian Tissues.: 20 normal ovarian tissue specimens are used as controls. These cases are treated by anti P16 antibody( p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267) , 1:500 concentration, over night duration and then treated by DAP secondary antibody.
Period: Overall Study
Arm/Group | IHC of P16 Expression in Malignant Ovarian Germ Cell Tumors. | IHC of P16 Expression in Benign Ovarian Germ Cell Tumors ( Mature Cystic Teratomas). | IHC of P16 Expression in Normal Ovarian Tissues.
Started | 22 | 20 | 20
Completed | 22 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Malignant Ovarian Germ Cell Tumors ( MOGCTs).: 22 cases of malignant ovarian germ cell tumors ; include Dysgerminoma , yolk sac tumor and immature teratomas will be treated by anti P16 antibody .
  p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267): Treatment of slides that cut from paraffin embedded blocks related to groups by immunohistochemical method by p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267).
- Normally Apparent Ovaries.: 20cases of normally apparent ovaries will be treated by anti P16 antibody .
- Total: Total of all reporting groups
Arm/Group | Malignant Ovarian Germ Cell Tumors ( MOGCTs). | Mature Cystic Teratomas. | Normally Apparent Ovaries. | Total
Number analyzed (Participants) | 22 | 20 | 20 | 62
Age, Continuous [Median (Full Range); unit: years] | 16.5 [12 to 23] | 31.5 [14 to 50] | 50 [42 to 64] | 30 [12 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 20 | 62
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 20 | 20 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 22 | 20 | 20 | 62
P16 cytoplasmic expression [Median (Full Range); unit: units on a scale] — Percentage of positive cells and the location of positive signals (nuclear or cytoplasmic) visually estimated for of lesions.
  German Semi-quantitative scoring system is used to evaluate P16 expression. A score according to the intensity of staining (no staining = 0, weak = 1, moderate = 2, strong= 3) And the extent of stained cells (0% = 0, 1-10% = 1, 11-50% =2, 51-80% = 3, 81-100% = 4).
  The final score will be determined by multiplying the intensity scores with the extent of positivity scores of stained cells, with the minimum score of 0 and a maximum score of 12.
  units on a scale | 7 [0 to 8] | 4 [0 to 6] | 0 [0 to 4] | 6 [0 to 8]
P16 nuclear expression [Median (Full Range); unit: units on a scale] — Percentage of positive cells and the location of positive signals (nuclear or cytoplasmic) visually estimated for of lesions.
  German Semi-quantitative scoring system is used to evaluate P16 expression. A score according to the intensity of staining (no staining = 0, weak = 1, moderate = 2, strong= 3) And the extent of stained cells (0% = 0, 1-10% = 1, 11-50% =2, 51-80% = 3, 81-100% = 4).
  The final score will be determined by multiplying the intensity scores with the extent of positivity scores of stained cells, with the minimum score of 0 and a maximum score of 12.
  units on a scale | 6 [0 to 8] | 4 [0 to 5] | 0 [0 to 3] | 4 [0 to 8]

OUTCOME MEASURES:

1. Primary Outcome: P16 Evaluation in Ovarian Germ Cell Tumors
Description: For P16 IHC staining, the percentage of P16 positive cells and the location of positive signals (nuclear or cytoplasmic) were visually estimated for neoplastic components of all lesions. German Semi-quantitative scoring system were used to evaluate P16 expression as every tumor will be given a score according to the intensity of the cytoplasmic and nucleic staining (no staining = 0, weak staining = 1, moderate staining = 2, strong staining = 3) And the extent of stained cells (0% = 0, 1-10% = 1, 11-50% =2, 51-80% = 3, 81-100% = 4). The final immunoreactive score will be determined by multiplying the intensity scores with the extent of positivity scores of stained cells, with the minimum score of 0 and a maximum score of 12 ( score 0, 1,2,3,4,6,8,9 and 12).
Time Frame: Antibody exposure overnight, assessed up to 3 days for each run of sections assessed.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Malignant Ovarian Germ Cell Tumors ( MOGCTs).: 22 cases of malignant ovarian germ cell tumors ; include Dysgerminoma , yolk sac tumor and immature teratomas will be treated by anti P16 antibody and Ki67 antibody.
  p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267): Treatment of slides that cut from paraffin embedded blocks related to groups by immunohistochemical method by p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267).Additional step for malignant cases , sections were treated by Ki67 antibody.
- Mature Cystic Teratomas.: 20 cases of mature teratomas will be treated by anti P16 antibody .
  p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267): Treatment of slides that cut from paraffin embedded blocks related to groups by immunohistochemical method by p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267).Additional step for malignant cases , sections were treated by Ki67 antibody.
- Normally Apparent Ovaries.: 20 cases of normally apparent ovaries will be treated by anti P16 antibody .
  p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267): Treatment of slides that cut from paraffin embedded blocks related to groups by immunohistochemical method by p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267).Additional step for malignant cases , sections were treated by Ki67 antibody.
Arm/Group | Malignant Ovarian Germ Cell Tumors ( MOGCTs). | Mature Cystic Teratomas. | Normally Apparent Ovaries.
Number analyzed (Participants) | 22 | 20 | 20
units on a scale
  P16 cytoplasmic expression | 7 [0 to 8] | 4 [0 to 6] | 0 [0 to 4]
  P16 nuclear expression | 6 [0 to 8] | 4 [0 to 5] | 0 [0 to 3]
Statistical Analysis 1: Comparison: Malignant Ovarian Germ Cell Tumors ( MOGCTs). vs Mature Cystic Teratomas. vs Normally Apparent Ovaries; Assessment of statistical differences in P16 expression between 3 groups. The immunohistochemical evaluation is done using German- semiquantitative scoring system. The score ranges from ( 0, 1,2,3,4,6,8,9 and 12). The data will entered on SPSS,version 24 as numbers. The test of significance is Kruskal Wallis was used to examine the Difference in Median between groups. Post-hoc test with Bonferroni Correction was used for Pairwise comparisons . A p-value < 0.05 was considered significant; Test type: Superiority; p = 0.001, Kruskal-Wallis — The test of significance is Kruskal Wallis was used to examine the Difference in Median between groups. Post-hoc test with Bonferroni Correction was used for Pairwise comparisons . A p-value < 0.05 was considered significant; Median Difference (Final Values) = 0.001, 95% CI 2-sided [0 to 8], Standard Deviation 1.5

2. Primary Outcome: Measurement of Ki67 Expression in Malignant Ovarian Germ Cell Tumors.
Description: For KI67 IHC staining for malignant cases, percentage of nuclear positivity stained cells were assessed, regardless intensity of staining in all sections examined (at least 1000 tumor cells were counted per section for estimation of KI index).Correlation analysis was used to test the association between Ki-67 and other variables (Spearman' Ranked correlation). A p-value < 0.05 was considered significant.
Time Frame: Antibody exposure 2 hrs , assessed up to 1 day for each run of sections assessed.
Population: Measurement of Ki67 expression in malignant ovarian germ cell tumors only. That explains why analysis obtained on Arm/Group 1 ( MOGCTs) only.
Measure: Median (Full Range); unit: percentage of Ki67 positive nuclear cell
Groups:
- Measurement of Ki67 Expression in Malignant Ovarian Germ Cell Tumors.: 22 cases of malignant ovarian germ cell tumors ; 5cases of dysgerminoma ( one of them is bilateral) , 9 cases of yolk sac tumor and 8 cases of immature teratoma.
  For KI67 IHC staining for malignant cases, percentage of nuclear positivity stained cells were assessed. KI67 LI is estimated by percentage of positive nuclei to all tumor cells from 0 to 100% scale.
Arm/Group | Measurement of Ki67 Expression in Malignant Ovarian Germ Cell Tumors.
Number analyzed (Participants) | 22
percentage of Ki67 positive nuclear cell | 15 [0 to 100]
Statistical Analysis 1: Comparison: Measurement of Ki67 Expression in Malignant Ovarian Germ Cell Tumors; Correlation between Ki 67 expression using percentage of Ki67 positive nuclei and P16 cytoplasmic expression using German semi quantitative score among MOGCT group. Data were analysed using IBM-SPSS version 24. Correlation analysis was used (Spearman' Ranked correlation, 2-tailed). A p-value < 0.05 was considered significant; Test type: Superiority; p = 0.009, Spearman's rank correlation coefficient( — Data were analysed using IBM-SPSS version 24. Correlation analysis was used (Spearman' Ranked correlation, 2-tailed). A p-value < 0.05 was considered significant; Hazard Ratio, log = 0.009, 95% CI 2-sided [0 to 8]

3. Secondary Outcome: Correlation Between P16 Cytoplasmic Score and FIGO Staging of MOGCTs.
Description: P16 cytoplasmic score is assessed by German quantitative scoring system by multiplying scores of intensity of staining ( 0= No , 1= weak , 2= moderate , 3 = strong ) in scores of intensity of staining ( 0 = less than 10% , 1= 11- 20 % , 2= 21-50 % , 3= 51-80% , 4= more than 80%) to induce final scores range between ( 0, 1,2,4,6,8,9 and 12).
  FIGO staging system for ovarian tumors between Stage I ( limited to ovaries) , II ( with pelvic extension) , III ( with peritoneal extension) and IV ( distant metastasis) , and it is reported from medical records of patients.
  One-way ANOVA was used to examine the Difference in Mean between groups. Post-hoc test with Bonferroni Correction was used for Pairwise comparisons . Data was expressed as mean (SD). A p-value < 0.05 was considered significant.
Time Frame: After obtaining of results and collecting raw data , within 2 months.
Population: P16 cytoplasmic score is assessed by German quantitative scoring system by multiplying scores of intensity of staining ( 0= No , 1= weak , 2= moderate , 3 = strong ) in scores of intensity of staining ( 0 = less than 10% , 1= 11- 20 % , 2= 21-50 % , 3= 51-80% , 4= more than 80%) to induce final scores range between ( 0, 1,2,4,6,8,9 and 12). FIGO staging for (malignant ovarian tumors only) is reported from medical records of patients . That explains why this measurement Arm/group 1( MOGCTs)only.
Measure: Mean (80% Confidence Interval); unit: score on a scale
Groups:
- Malignant Ovarian Germ Cell Tumors ( MOGCTs).: 22 cases of malignant ovarian germ cell tumors ; include Dysgerminoma , yolk sac tumor and immature teratomas will be treated by anti P16 antibody
Arm/Group | Malignant Ovarian Germ Cell Tumors ( MOGCTs).
Number analyzed (Participants) | 22
score on a scale | 11 [9.5 to 13.5]
Statistical Analysis 1: Comparison: Malignant Ovarian Germ Cell Tumors ( MOGCTs); Correlation between P16 cytoplasmic score using German semi-quantitative system and FIGO staging of MOGCTs was done via One-way ANOVA was used to examine the Difference in Mean between groups. Post-hoc test with Bonferroni Correction was used for Pairwise comparisons .Data was expressed as mean (SD); Test type: Superiority — One-way ANOVA was used to examine the Difference in Mean between groups. Post-hoc test with Bonferroni Correction was used for Pairwise comparisons .Data was expressed as mean (SD). P value is significant if less than 0.05; p = 0.699, ANOVA — One-way ANOVA was used to examine the Difference in Mean between groups. Post-hoc test with Bonferroni Correction was used for Pairwise comparisons .Data was expressed as mean (SD). P value is significant if less than 0.05; Mean Difference (Final Values) = 11, 80% CI 2-sided [9.5 to 13], Standard Deviation 1.5

ADVERSE EVENTS:
Time Frame: 1 year
Description: Nature of specimen is paraffin embedded tissue blocks , therefore there is no mortality , harm or serious Adverse Events were obtained to the participants. This explained why "0" is a total number of Participants at Risk.
Groups:
- Immunohistochemical Expression of P16 Expression in Malignant Ovarian Germ Cell Tumors.: 22cases of malignant ovarian germ cell tumors ; 5 cases of dysgerminoma ( one of them is bilateral) , 9cases of yolk sac tumor and 8 cases of immature teratoma. These cases are treated by anti P16 antibody( p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267) , 1:500 concentration, over night duration and then treated by DAP secondary antibody . Finally assessed by visualized peroxidase method.
- Immunohistochemical Expression of P16 Expression in Benign Ovarian Germ Cell (MCTs): 20 cases of mature cystic teratomas ; were treated by anti P16 antibody( p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267) , 1:500 concentration, over night duration and then treated by DAP secondary antibody . Finally assessed by visualized peroxidase method.
- Immunohistochemical Expression of P16 Expression in Normal Ovarian Tissues.: 20 cases of normal ovarian tissues were treated by anti P16 antibody( p16INK4a Recombinant Rabbit Monoclonal Antibody (RM267) , 1:500 concentration, over night duration and then treated by DAP secondary antibody . Finally assessed by visualized peroxidase method.
Arm/Group | Immunohistochemical Expression of P16 Expression in Malignant Ovarian Germ Cell Tumors. | Immunohistochemical Expression of P16 Expression in Benign Ovarian Germ Cell (MCTs) | Immunohistochemical Expression of P16 Expression in Normal Ovarian Tissues.
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT04283773/Prot_SAP_ICF_000.pdf